CLINICAL TRIAL: NCT06235320
Title: Paracetamol Impact Study: Prostaglandin Synthesis and Blood Pressure Effects (PIS-PaB)
Brief Title: Paracetamol Effect on Prostaglandins and Blood Pressure
Acronym: PIS-PaB
Status: Not yet recruiting | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Engi Algharably, Dr., Charite University, Berlin, Germany
Other Study IDs: PIS-PaB
Record Dates: First submitted 2024-01-18; First posted 2024-01-31 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Paracetamol group
  Interventions: Other: routine clinical treatment of pain with paracetamol or ibuprofen
- Ibuprofen group
  Interventions: Other: routine clinical treatment of pain with paracetamol or ibuprofen

INTERVENTIONS:
Other: routine clinical treatment of pain with paracetamol or ibuprofen — No intervention beside clinical routine management

SUMMARY:
This research program aims to investigate the influence of paracetamol on blood pressure and the cyclooxygenase (COX) - prostaglandine (PG) pathway in patients with pain. Through an observational pilot study, we will use advanced LC/ESI-MS/MS methodology to analyze the COX-OG pathway in plasma and urine. The study will assess the effects of paracetamol compared to ibuprofen, considering different types of pain. The primary focus is to understand the changes in blood pressure and the COX-PG pathway upon initiation or discontinuation of paracetamol, with safety analysis as a secondary consideration.

ELIGIBILITY:
Inclusion Criteria:

* Headache and orosurgical patients treated at the respective charite outpatient clinic.
* Age 18 years or older
* Able to consent
* Patients with migraine type headache treated with paracetamol or ibuprofen within the last 12 hours or not treated with paracetamol or ibuprofen within the last 48 hours
* Patients treated with with paracetamol or ibuprofen undergoing orosurgery for wisedome tooth extraction

Exclusion Criteria:

* Pregnancy
* Arterial hypertension
* Use of beta blockers
* Use of COX inhibitors other than paracetamol or ibuprofen, including low-dose acetylsalicylic acid
* Stable prophylactic therapy of migraine for less than 3 weeks
* Use of tryptans in the last two days (Frovatriptane in the last 6 days)
* Oral surgery patients using paracetamol or ibuprofen in the last 24 hours
* Known allergy to paracetamol or ibuprofen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The first cohort consists of patients of the headache consultation at Charité Campus Mitte, where data is collected both within and outside of clinical routine, whereby the medical care of the respective patients takes place in the usual routine.
  The second cohort consists of patients attending oral surgery consultations at the Institute of Dentistry, Oral and Maxillofacial Surgery, for whom data is also collected both within and outside of clinical routine, whereby the medical care of the respective patients takes place in the usual routine.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Prostanoid levels | just before treatment and 24 hours after treatment with paracetamol or ibuprofen
  A comprehensive lipidomic analysis measuring the levels of prostanoids in plasma and spot urine samples using liquid chromatography tandem mass spectrometry (LC/ESI-MS/MS) technology in all participants.

SECONDARY OUTCOMES:
Blood pressure | just before treatment and 24 hours after treatment with paracetamol or ibuprofen
  Automated office and ambulatory blood pressure measurement

IPD SHARING:
Plan to Share IPD: No
No plan to share individual patient data